CLINICAL TRIAL: NCT04394481
Title: Extension of the Analgesia of an Interscalene Block of the Brachial Plexus by Combined Injection of Dexamethasone and Dexmedetomidine, After Arthroscopic Shoulder Surgery: Randomized, Controlled, Double-blind Trial
Brief Title: Extension of Analgesia by Combined Injection of Dexamethasone and Dexmedetomidine After Arthroscopic Shoulder Surgery
Acronym: INDEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-000611-74
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Ropivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DMD (Experimental): Ropivacaine: perinervous injection (interscalene block) Dexamethasone: IV injection Dexmedetomidine: IV injection (1µg/kg)
  Interventions: Drug: Dexmedetomidine; Drug: Ropivacaine; Drug: Dexamethasone
- Control (Active Comparator): Ropivacaine: perinervous injection (interscalene block) Dexamethasone: IV injection
  Interventions: Drug: Ropivacaine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexmedetomidine — IV injection (1 µg/kg - 100 mL) before anesthetic induction
  Arms: DMD
Drug: Ropivacaine — Perinervous injection between C5 and C6 nerve roots / interscalene block (0.75% - 20 mL)
Drug: Dexamethasone — IV injection (0.15 mg/kg) during anesthetic induction

SUMMARY:
The main objective of the study is to demonstrate the efficacy of Dexmedetomidine on the prolongation of analgesia obtained by interscalenic bloc of the brachial plexus and intravenous injection of Dexamethasone (efficacy objective).

DETAILED DESCRIPTION:
This is an interventional, comparative, randomized, controlled study versus reference treatment, in 2 parallel groups, double blind (patient and evaluator), multicenter, aiming to demonstrate the superiority of This is an interventional, comparative, randomized, controlled study versus reference treatment, in 2 parallel groups, double blind (patient and evaluator), multicenter, aiming to demonstrate the superiority of Dexmedetomidine over the absence of Dexmedetomidine, in adjuvantation of a loco regional anesthesia (interscalenic bloc of the brachial plexus + intravenous injection of Dexamethasone), on the prolongation of the analgesia, following a surgery of the rotator cuff of the shoulder under arthroscopy.

Patients will be randomized into 2 groups according to the treatment received:

* Dexmedetomidine;
* Nothing (control arm). The investigator (anesthesiologist) who will perform the randomization will not be blinded to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patient undergoing arthroscopic shoulder surgery to repair the rotator cuff tendons;
* Patient capable of understanding the information related to the study, of reading the information leaflet and agreeing to sign the consent form.

Exclusion Criteria:

* Patient on oral morphines before surgery;
* Contraindication to performing a general anesthesia associated with a shoulder loco regional anesthesia in a single injection;
* Contraindication to take oral morphines;
* Any non-arthroscopic repair (intraoperative conversion to "open sky" technique);
* Any other loco regional anesthesia than an interscalenic block (change of intraoperative strategy);
* Pregnant or lactating woman;
* Intolerance or allergy or contraindication to one of the treatments under study;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
Effectiveness of dexmedetomidine in prolonging analgesia | 96 hours
  Delay between the start of the loco regional anesthésia (Hour 0) and the first post-operative oral morphine intake.

SECONDARY OUTCOMES:
Duration of the motor block | 96 hours
  Delay between Hour 0 (H0) and the moment when the patient can move his/her forearm and / or his/her arm again
Duration of the sensitive block | 96 hours
  Delay between H0 and the moment when the patient claims to have started to experience paraesthesia on his/her shoulder after the operation
Numerical scale from 0 to 10 | 48 hours
  Pain scores at rest and in motion estimated by the patient at Hour 4 (H4), Hour 12 (H12), Hour 24 (H24) and Hour 48 (H48)
Oral opioid analgesics | 48 hours
  Cumulative amount of oral opioid analgesics taken during the 48 hours post-operative
Safety analysis | 96 hours
  Evaluation of adverse events
4-level Likert scale | 96 hours
  Patient satisfaction with regard to analgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Julien CABATON, Principal Investigator — Scientific Committee
Locations (1):
- Hôpital privé jean Mermoz, Lyon, France

IPD SHARING:
Plan to Share IPD: No